CLINICAL TRIAL: NCT02137304
Title: A Method to Optimize Mecanical In-exsufflation in Neuromuscular Diseases
Acronym: COUGHELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01771-44
Record Dates: First submitted 2014-04-17; First posted 2014-05-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-11

CONDITIONS: Neuromuscular Disease
Keywords: cough help; in-exsufflation; neuromuscular disease; cough assistance optimization; efficient cough flow
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuromuscular patients (Experimental): Cough Assist® (JH Emerson Compagny, Cambridge, MA, USA)
  Interventions: Device: Cough Assist® (JH Emerson Compagny, Cambridge, MA, USA)

INTERVENTIONS:
Device: Cough Assist® (JH Emerson Compagny, Cambridge, MA, USA) — Cough Assist® (JH Emerson Compagny, Cambridge, MA, USA) mechanical insufflation to increase peak cough flow

SUMMARY:
The investigators want to demonstrate that there is an optimal expiratory pressure when using mecanical in-exsufflation for each patient in neuromuscular disease. This compromise is between the need to generate a high pressure difference between alveoli and the mouth and the need to avoide and superior airways collapsus.

DETAILED DESCRIPTION:
he investigators want to demonstrate that there is an optimal expiratory pressure when using mecanical in-exsufflation for each patient in neuromuscular disease. This compromise is between the need to generate a high pressure difference between alveoli and the mouth and the need to avoide and superior airways collapsus.

ELIGIBILITY:
Inclusion Criteria:

* man or female age18 years
* neuromuscular disease
* coughassist adaptation treatment
* peak cough flow<270liter/minute

Exclusion Criteria:

* acute organ failure
* insufflation contrindication
* pregnant women/no affiliation to a social security scheme
* plan of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
optimal negative pressure treshold value | 20 minutes
  Optimal negative pressure treshold value measured for a flow superior or equal to 160 liter/minute and 270 liter/minute

SECONDARY OUTCOMES:
optimal pressure treshold based on the best peak flow. | 10 minutes
volume-flow curve aspect | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frederic LOFASO, Pr, Principal Investigator — AP-HP Hopital R. Poincaré Garches
Locations (1):
- Hôpital R. POINCARE, Garches, France

REFERENCES:
- [Derived] Lacombe M, Bore A, Amo Castrillo LD, Boussaid G, Falaize L, Vlachos E, Orlikowski D, Prigent H, Lofaso F. Peak Cough Flow Fails to Detect Upper Airway Collapse During Negative Pressure Titration for Cough-Assist. Arch Phys Med Rehabil. 2019 Dec;100(12):2346-2353. doi: 10.1016/j.apmr.2019.06.012. Epub 2019 Jul 24. PMID 31351076